CLINICAL TRIAL: NCT02197117
Title: Effect of Remote Ischaemic Conditioning in STEMI Patients Treated by thromboLYSIS: A Randomised Controlled Clinical Trial (the ERIC-LYSIS Study)
Brief Title: Effect of Remote Ischemic Conditioning in Heart Attack Patients
Acronym: ERIC-LYSIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Principal Investigator, Derek Hausenloy, Professor in Cardiovascular Medicine, University College, London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ERIC-LYSIS
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: ST-segment elevation myocardial infarction (STEMI); thrombolysis, remote ischemic conditioning, myocardial infarct size, cardioprotection
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remote ischemic conditioning (Active Comparator): Standard blood pressure cuff placed on upper arm and inflated to 200 mmHg. The cuff is left inflated at this level for 5 minutes and then rapidly deflated to 0 mmHg left deflated for 5 minutes0 this cycle is repeated 4 times in total.
  Interventions: Device: Remote ischemic conditioning
- Control (Sham Comparator): Standard blood pressure cuff placed on upper arm and left un-inflated for 40 minutes, and then cuff is removed.
  Interventions: Device: Control

INTERVENTIONS:
Device: Remote ischemic conditioning
  Arms: Remote ischemic conditioning
Device: Control
  Arms: Control

SUMMARY:
New treatments are required to improve health outcomes in patients with ischemic heart disease. This is especially so in developing countries such as Mauritius in which optimal therapy for acute myocardial infarction may not be widely available. For example for patients presenting with a heart attack (caused by a blockage in one of the heart blood vessels) the treatment of choice would be to remove the blockage by primary percutaneous coronary intervention (PCI) using an angioplasty balloon and put a stent (a spring-like structure) to keep the artery opened. However, PCI is not widely available in Mauritius and heart attack patients are given clot-busting therapy to remove the blockage, but this is not as effective as PCI.

Therefore, in this research study we investigate a new cheap treatment that may help protect the heart against damage during a heart attack, called remote ischemic conditioning (RIC), in which a blood pressure cuff is placed on the upper arm and inflated for 5 minute and deflated for 5 minutes a cycle which is repeated 4 times in total in patients presenting with a heart attack. By temporarily depriving oxygen and nutrients to the arm with the blood pressure cuff a protective signal can be relayed to the heart to reduce the amount of damage occurring during the heart attack and thereby prevent the onset of heart failure.

Study hypothesis: Remote ischaemic conditioning will reduce the amount of damage occurring to the heart muscle during a heart attack..

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Presentation within 12 hours of onset of chest pain
* ECG showing ST-segment elevation of ≥0.1mV in two contiguous leads (≥0.2mV in leads V1-V3)

Exclusion Criteria:

-None -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2011-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Myocardial infarct size | Measured by 24 hr area under the curve serum CK-MB and Troponin-T sampled a time 0, 6, 12, and 24 hrs post-thrombolysis
  Measured by 24 hr area under the curve serum CK-MB and Troponin-T sampled a time 0, 6, 12, and 24 hrs post-thrombolysis.

SECONDARY OUTCOMES:
Acute kidney injury | Measured by serum creatinine at 24 hours
  Measured by serum creatinine at 24 hours.

CONTACTS AND LOCATIONS:
Locations (5):
- Mauritius (5):
  - Victoria Hospital, Candos
  - Flacq Hospital, Centre de Flacq
  - Sir Seewoosagur Ramgoolam National Hospital, Pamplemousses
  - Dr AG Jeetoo Hospital, Port Louis
  - Jawaharlal Nehru Hospital, Rose Belle